CLINICAL TRIAL: NCT04394208
Title: Trial of Silymarin in Adults With COVID-19 Pneumonia
Brief Title: Silymarin in COVID-19 Pneumonia
Acronym: SCOPE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Mohammed Korany Salem, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU COVID-19 Study Group
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; Viral Pneumonia Human Coronavirus
Keywords: COVID-19; SARS-CoV-2; Viral Pneumonia; Drug; Silymarin; Treatment; p38 MAPK Inhibitor
MeSH Terms: conditions — COVID-19; Pneumonia, Viral | interventions — Silymarin

STUDY DESIGN:
Intervention Model Description: Group 1 (Control): Includes 25 patients with COVID-19 pneumonia receiving standard of care as per Ministry of Health Protocol of Treatment + placebo Group 2 (Intervention): Includes 25 patients with COVID-19 pneumonia receiving standard of care as per Ministry of Health Protocol of Treatment + Silymarin Oral at a dose of 420 mg/day in 3 divided doses.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Placebo Comparator): Patients with COVID-19 pneumonia receiving standard of care as per Ministry of Health Protocol of Treatment plus placebo
  Interventions: Drug: Placebo
- Group 2 (Experimental): patients with COVID-19 pneumonia receiving standard of care as per Ministry of Health Protocol of Treatment + Silymarin Oral 420mg/day in 3 divided doses
  Interventions: Drug: Silymarin

INTERVENTIONS:
Drug: Silymarin — Silymarin Oral at a dose of 420 mg/day in 3 divided doses.
  Arms: Group 2
Drug: Placebo — Placebo comparator
  Arms: Group 1

SUMMARY:
A randomized placebo controlled trial to assess the clinical outcome in COVID-19 Pneumonia following administration of Silymarin owing to its role as a p38 MAPK pathway inhibitor and its antiviral, anti-inflammatory and anti-oxidant effects

DETAILED DESCRIPTION:
To date, there are no drugs or other therapeutics approved by the U.S. Food and Drug Administration (FDA) to prevent or treat COVID-19 that has spread globally resulting in the ongoing pandemic as declared by the World Health Organization (WHO) on 11 March 2020. While the majority of patients have mild symptoms, some progress to viral pneumonia and multi-organ failure (MOF).

Older age, cardiovascular disease, diabetes mellitus, chronic respiratory illness, systemic hypertension, and malignancy are all associated with an increased risk of death in COVID-19.

In fatal cases of human severe acute respiratory syndrome-associated coronavirus (SARS-CoV), Middle East respiratory syndrome coronavirus (MERS-CoV) and SARS-CoV-2 infections, patients suffer from severe respiratory distress necessitating mechanical ventilation. Previous studies showed that genetic susceptibility and inflammatory cytokines (Interleukins: IL-6, 8, 10, Tumor Necrosis Factor [TNF] and Vascular endothelial growth factor [VEGF]) are closely related to the occurrence of acute respiratory distress syndrome (ARDS).

Cytokine storm is another life-threatening condition, and likely a leading cause of fatality.

Rapid viral replication and apoptosis together with virus-induced angiotensin-converting enzyme 2 (ACE-2) down-regulation and shedding and antibody-dependent enhancement (ADE) are responsible for aggressive inflammation caused by SARS-CoV-2, which is closely related to SARS-CoV; where both viruses hijack the same entry receptor ACE-2 suggesting the likelihood of the same population of cells being targeted and infected.

A Previous study demonstrated that p38 mitogen-activated protein kinase (p38 MAPK) and its downstream targets are activated in SARS-CoV infected Vero E6 cells and that activation of p38 MAPK enhances the cytopathic effects of SARS-CoV infection.

Interestingly, the p38 MAPK pathway is a key regulator of proinflammatory cytokine synthesis, which may contribute to the chronic low-grade inflammation observed with ageing. Another study hypothesized that ageing up-regulates the activation of p38 MAPK as well as the pro-inflammatory cytokines TNF-α, IL-1β and IL-6 in mouse lung and is accompanied by disturbances in oxidant-antioxidant status.

Furthermore, it was shown that p38 MAPK pathway is involved in the inflammatory response induced by cigarette smoke exposure, endotoxin and oxidative stress, through activation and release of pro-inflammatory cytokines, and it was postulated that inhibition of p38 MAPK prevented allergen-induced pulmonary eosinophilia, mucus hypersecretion and airway hyper-responsiveness.

p38 MAPK was identified as a possible target in vascular cells, which can be activated by high glucose levels and diabetes, where at moderate and commonly encountered levels of hyperglycemia, p38 MAPK appears to be activated by PKC-δ isoform-dependent processes.

Numerous preclinical studies have addressed the role of p38 MAPK in ischemic heart disease, myocardial infarction, and atherosclerosis.

Hence, The investigators of this clinical trial have concluded that p38 MAPK pathway activation could explain the increased risk of death from COVID-19 in older age, diabetes mellitus, cardiovascular disease, systemic hypertension and chronic respiratory diseases. Therefore, p38 MAPK inhibitors may play a promising role in the treatment of SARS-CoV-2 and COVID-19 improving the clinical outcomes.

Silymarin, an extract from the seed of the milk thistle plant (Silybum marianum [S. marianum]) is widely known for its hepatoprotective functions, mainly due to its anti-oxidative, anti-inflammatory, and immunomodulatory effects.

Recent studies documented the antiviral activities of Silymarin against several viruses; including flaviviruses (hepatitis C virus and dengue virus), togaviruses (Chikungunia virus and Mayaro virus), influenza virus, hepatitis B virus and Human Immunodeficiency Virus (HIV); in addition to its anti-oxidative and anti-inflammatory role.

Furthermore, a recent study demonstrated the role of Silymarin in attenuating cigarette smoke extract-induced inflammation via simultaneous inhibition of autophagy and extracellular signal-regulated kinase/p38 mitogen-activated protein kinase (ERK/ p38 MAPK) pathway in human bronchial epithelial cells, as well as attenuating up-regulation of pro-inflammatory cytokines TNF-α, IL-6 and IL-8 and concluded that Silymarin might be an ideal agent treating inflammatory pulmonary diseases.

This clinical trial aim at evaluating the role of Silymarin in the treatment of adults with COVID-19 Pneumonia

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients with CT Chest-proven viral pneumonia with any degree of severity.

Exclusion Criteria:

* Patients < 18 years of age.
* Patients with mild symptoms (as per WHO criteria) of SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-16 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | 7-28 days
  Defined as the time from randomization to an improvement of two points (from the status of randomization) on seven category ordinal scale or live discharge from the hospital, whichever comes first.

SECONDARY OUTCOMES:
Clinical outcome | 7-14 days
  Clinical status as assessed with the seven-category ordinal scale on days 7 and 14
Duration of Mechanical Ventilation | Randomization till hospital discharge or death whichever came first, assessed up to 28 days
  Time in days patient was intubated
Hospitalization | Randomization till hospital discharge or death whichever came first, assessed up to 28 days
  Total days of hospitalization
Virologic Response | Randomization till discharge, up to 28 days
  number of days patient remained with positive RT-PCR SARS-CoV-2 swab
Adverse events | Randomization till hospital discharge, up to 28 days
  Any adverse events whether related to medication or not

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Liu CH, Jassey A, Hsu HY, Lin LT. Antiviral Activities of Silymarin and Derivatives. Molecules. 2019 Apr 19;24(8):1552. doi: 10.3390/molecules24081552. PMID 31010179
- [Background] Li D, Hu J, Wang T, Zhang X, Liu L, Wang H, Wu Y, Xu D, Wen F. Silymarin attenuates cigarette smoke extract-induced inflammation via simultaneous inhibition of autophagy and ERK/p38 MAPK pathway in human bronchial epithelial cells. Sci Rep. 2016 Nov 22;6:37751. doi: 10.1038/srep37751. PMID 27874084